CLINICAL TRIAL: NCT03670732
Title: Nasal Intermittent Positive Pressure Ventilation vs. Nasal Continuous Positive Airway Pressure at Equivalent Mean Airway Pressure in Preterm Infants: Effect on Oxygenation, CO2 Elimination, Work of Breathing and Frequency of Cardio-respiratory Events.
Brief Title: CPAP vs.Unsynchronized NIPPV at Equal Mean Airway Pressure
Acronym: NICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain needed equipment and COVID-related suspension of clinical research
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Martin Keszler, Professor of Pediatrics, Associate Director of NICU, Director of Respiratory Care, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1010049; WIH 17-0037 (Other: Women and Infants Hospital of Rhode Island)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Prematurity; Respiratory Distress Syndrome; Apnea of Prematurity
Keywords: Continuous positive airway pressure; Nasal intermittent positive pressure ventilation; Mean airway pressure; Apnea; Bradycardia; Prematurity
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Apnea; Bradycardia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Crossover non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP first (Active Comparator): The intervention is application of continuous positive airway pressure (CPAP). The order of the two interventions of this crossover study is randomized but each subject will be exposed to both interventions. The period of CPAP will be compared to the period of NIPPV.
  Interventions: Other: continuous positive airway pressure; Other: nasal intermittent positive pressure ventilation
- NIPPV first (Active Comparator): The intervention is application of nasal intermittent positive pressure ventilation (NIPPV). The order of the two interventions of this crossover study is randomized but each subject will be exposed to both interventions. The period of CPAP will be compared to the period of NIPPV.
  Interventions: Other: continuous positive airway pressure; Other: nasal intermittent positive pressure ventilation

INTERVENTIONS:
Other: continuous positive airway pressure — Continuous positive airway pressure is applied for 12 hours at a mean airway pressure that is the same as the subject was receiving prior to entry into the study
  Other Names: CPAP
Other: nasal intermittent positive pressure ventilation — NIPPV is applied for 12 hours at a mean airway pressure that is the same as the subject was receiving prior to entry into the study
  Other Names: NIPPV

SUMMARY:
This study seeks to determine if standard continuous positive airway pressure, known as CPAP is as effective as a more complicated approach that generates intermittent increases in airway pressure applied to the nostrils via a breathing machine. The latter is known as NIPPV and requires costly equipment to operate. Previous studies did not ensure that the average pressure applied to the lungs was equal and thus did not make for a fair comparison. The investigators believe that when the same average pressure is applied with the two techniques, CPAP is just as effective as NIPPV and may have fewer side effects, such as blowing air into the stomach. Each baby will receive CPAP or NIPPV in a random sequence for a period of 12 hours, followed by 12 hours on the alternate technique.

DETAILED DESCRIPTION:
This is a pilot clinical trial to evaluate the comparative effectiveness of two commonly used types of non-invasive respiratory support. Preterm infants < 34 weeks gestational age, who are stable on either of the two modalities of support will be studied in a cross-over study design, such that each subject acts as his/her own control. The study will assess the relative efficacy of these modalities when used with equal mean airway pressure comparing measures of oxygenation, CO2 removal, apnea/bradycardia/desaturation events and work of breathing. The initial phase of the study is complete and preliminary analysis supports the hypothesis that there is no difference between the modalities when the mean airway pressure is equal. However we recognized that use of the RAM cannula, which does not transmit pressure effectively is an important study limitation. The findings are valid, but may only be applicable to this interface, which is widely used, but increasingly recognized as flawed. We are now extending the study to determine if the findings will be the same when short bi-nasal prongs are used.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age 23-34 completed weeks
* Stable on non- invasive respiratory support for at least 24h
* CPAP level of 7-12 cmH2O or NIPPV with MAP 7-12 cmH2O
* FiO2 requirement of <0.40

Exclusion Criteria:

* Clinical instability as judged by the clinical team
* FiO2 requirement of > 0.40 for more than 60 min.
* >10 apnea/bradycardia/desaturation events in past 24 h requiring moderate or vigorous stimulation.
* Anticipated intubation within next 24 h.
* Active abdominal pathology (Spontaneous Intestinal Perforation, confirmed or suspected Necrotizing Enterocolitis, bowel obstruction).
* Hemodynamically significant patent ductus arteriosus (PDA)
* Anticipated weaning off non-invasive support in the next 24 h.
* Any major congenital anomalies, congenital heart disease (other than PDA, atrial septal defect or ventricular septal defect) and cardiac arrhythmias
* Lack of study equipment or personnel
* Lack of parental consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Apnea/bradycardia events | Duration of intervention (12 hours)
  Number of episodes of apnea and/or bradycardia that trigger alarm on the bedside monitor

SECONDARY OUTCOMES:
Number of of desaturation events | Duration of intervention (12 hours)
  Number of episodes of pulse oximetry readings that trigger alarm on the bedside monitor
Mean oxygen saturation by pulse oximetry and proportion of time below 88% | Duration of intervention (12 hours)
  Mean oxygen saturation by pulse oximetry and proportion of time at saturation <88%
Mean transcutaneous PCO2 and proportion of time >55 torr | Duration of intervention (12 hours)
  Mean transcutaneous PCO2 and proportion of time at PCO2 > 55 torr
Mean fraction of inspired oxygen | Duration of intervention (12 hours)
  Mean fraction of inspired oxygen (FIO2)
Mean respiratory rate | Duration of intervention (12 hours)
  Mean respiratory rate
Mean degrees of phase lag by RIP | Duration of intervention (12 hours)
  Estimate of work of breathing based on phase angle as determined by respiratory inductive plethysmography
Number of episodes of feeding intolerance | Duration of intervention (12 hours)
  number of instances of interruption of feeding, abdominal radiographs
Instances of treatment failure | Duration of intervention (12 hours)
  Inability to tolerate assigned treatment by pre-defined criteria

CONTACTS AND LOCATIONS:
Overall Officials: Martin Keszler, MD, Principal Investigator — Brown University
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No